CLINICAL TRIAL: NCT02127983
Title: Engaging Informal Health Care Providers on Case Detection and Treatment Initiation Rates for TB and HIV in Rural Malawi (Triage Plus): a Cluster Randomised Health System Intervention Trial
Brief Title: Engaging Informal Health Care Providers on Case Detection and Treatment Initiation Rates for TB and HIV in Rural Malawi (Triage Plus)
Acronym: Triage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Research for Equity And Community Health REACH Trust (Unknown); Ministry of Health and Population, Malawi (Other Government); LHL International Tuberculosis Foundation (Unknown); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: TriagePlus
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2012-12

CONDITIONS: Tuberculosis; HIV
Keywords: TB, HIV, case finding, access, informal providers
MeSH Terms: conditions — Tuberculosis | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early intervention (Experimental): Early intervention arm engaging informal providers Received the intervention early in the first 12 months
  Interventions: Behavioral: Early intervention
- Delayed intervention (Active Comparator): Delayed intervention arm, engaging informal providers Received the intervention after one year
  Interventions: Behavioral: Delayed intervention

INTERVENTIONS:
Behavioral: Early intervention — Training non-paid informal healthcare providers (such as store-keepers) in TB and HIV disease recognition, sputum specimen collection, referral to the public health system, and raising community awareness.
  Front line public health personnel and community leaders were sensitised to support the intervention
  Other Names: Early intervention arm engaging informal providers; Received the intervention early in the first 12 months
  Arms: Early intervention
Behavioral: Delayed intervention — Delayed intervention arm, engaging informal providers Received the intervention after one year
  Arms: Delayed intervention

SUMMARY:
The intervention consisted of training non-paid informal healthcare providers (such as store-keepers) in TB and HIV disease recognition, sputum specimen collection, referral to the public health system, and raising community awareness. Front line public health personnel and community leaders were sensitised to support the intervention.

DETAILED DESCRIPTION:
A phased, matched, parallel cluster design was used to randomise three clusters (average population size per cluster = 200,714) to the Early intervention arm (received the intervention early in the first 12 months) and an equal number to the Delayed intervention arm (average population size per cluster = 209,564) which received the intervention after one year. Data for impact evaluation were obtained from routine patient registers in all the health facilities and patients were blindly allocated to the respective clusters based on residential address. Treatment initiation rates (expressed as incidence rate ratios) for TB and Anti Retroviral Therapy (ART) over the 12 months period were the primary outcome measures for each of the studied conditions. Poisson regression models with robust standard errors were used to assess the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* People accessing informal providers with possible TB or HIV

Exclusion Criteria:

* children
* people already with a diagnosis of TB or HIV

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200000 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
TB and HIV treatment initiation | 2 years
  the cumulative counts of patients initiating TB and HIV treatment per 10,000 adults aged 12 years and above each month over the intervention period

SECONDARY OUTCOMES:
TB and HIV diagnostic uptake rates. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Thomson, MSc, Principal Investigator — LSTM
Locations (1):
- REACH Trust, Lilongwe, Malawi

REFERENCES:
- [Derived] Bello G, Faragher B, Sanudi L, Namakhoma I, Banda H, Malmborg R, Thomson R, Squire SB. The effect of engaging unpaid informal providers on case detection and treatment initiation rates for TB and HIV in rural Malawi (Triage Plus): A cluster randomised health system intervention trial. PLoS One. 2017 Sep 6;12(9):e0183312. doi: 10.1371/journal.pone.0183312. eCollection 2017. PMID 28877245